CLINICAL TRIAL: NCT05895981
Title: An Exploratory Clinical Trial to Evaluate the Safety and Efficacy of Sacral Nerve Stimulation in Patients
Brief Title: Exploratory Clinical Trial of Safety and Efficacy of Sacral Nerve Stimulation in Patients With Ulcerative Colitis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20232100
Record Dates: First submitted 2023-05-15; First posted 2023-06-09 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-04

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; sacral nerve stimulation
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sacral nerve stimulation (Experimental)
  Interventions: Device: G132 system, Beijing PINS Medical Co., China

INTERVENTIONS:
Device: G132 system, Beijing PINS Medical Co., China — Neuromodulation was performed according to the usual protocol

SUMMARY:
Although the incidence of inflammatory bowel disease is stable in North American and European countries, the incidence of inflammatory bowel disease is increasing in newly industrialized countries, especially in China. The treatment drugs for ulcerative colitis include 5-aminosalicylic acid (5-ASA), glucocorticoids, immunosuppressants, and biological agents.

The aim of this exploratory Clinical Trial is to evaluate the safety and efficacy of sacral nerve stimulation in patients with ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* ulcerative colitis diagnosed for at least 3 mouths.
* Mayo score 6-12, Mayo endoscopic score 2-3 points
* resistant to medical treatment

Exclusion Criteria:

* Treatment-naive ulcerative colitis (no previous treatment)
* Acute severe ulcerative colitis
* Currently taking any biologicals
* Previous surgical treatment or severe colitis at imminent risk of surgery
* infective colitis
* Other systemic diseases
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Mayo score at week 12 | 12 weeks
  Mayo score at 12 week minus the Mayo score at baseline. The range of Mayo score is 0-12, and higher scores mean worse outcome.

SECONDARY OUTCOMES:
Change from baseline in the Mayo score at week 24, and 52 | 24 and 52 weeks
  Mayo score at 24 week minus the Mayo score at baseline. The range of Mayo score is 0-12, and higher scores mean worse outcome.
Clinical remission at Week 12, 24, and 52 | 12, 24, and 52 weeks
  overall score ≤2 [and no individual subscore >1]
Clinical response at Week 12, 24, and 52 | 12, 24, and 52 weeks
  defined as the reduction of baseline scores by ≥3 points
Change from baseline in the Truelove and Witts Severity Index at Week 12, 24, and 52 | 12, 24, and 52 weeks
  Truelove and Witts Severity Index
Endoscopic remission at Week 12, 24, and 52 | 12, 24, and 52 weeks
  defined as Mayo endoscopic score ≤ 1
Fecal calprotectin levels at baseline, week 4, 8, 12, 24 and 52 | baseline, 4, 8, 12, 24, and 52 weeks
  fecal sample
erythrocyte sedimentation rate levels at baseline, week 4, 8, 12, 24 and 52 | baseline, 4, 8, 12, 24, and 52 weeks
  blood sample
C reactive protein levels at baseline, week 4, 8, 12, 24 and 52 | baseline, 4, 8, 12, 24, and 52 weeks
  blood sample
pancreatic polypeptide levels at baseline, week 4, 8, 12, 24 and 52 | baseline, 4, 8, 12, 24, and 52 weeks
  blood sample
norepinephrine levels at baseline, week 4, 8, 12, 24 and 52 | baseline, 4, 8, 12, 24, and 52 weeks
  blood sample
interleukin-1β levels at baseline, week 4, 8, 12, 24 and 52 | baseline, 4, 8, 12, 24, and 52 weeks
  blood sample
interleukin-2 levels at baseline, week 4, 8, 12, 24 and 52 | baseline, 4, 8, 12, 24, and 52 weeks
  blood sample
interleukin-4 levels at baseline, week 4, 8, 12, 24 and 52 | baseline, 4, 8, 12, 24, and 52 weeks
  blood sample
interleukin-5 levels at baseline, week 4, 8, 12, 24 and 52 | baseline, 4, 8, 12, 24, and 52 weeks
  blood sample
interleukin-6 levels at baseline, week 4, 8, 12, 24 and 52 | baseline, 4, 8, 12, 24, and 52 weeks
  blood sample
interleukin-8 levels at baseline, week 4, 8, 12, 24 and 52 | baseline, 4, 8, 12, 24, and 52 weeks
  blood sample
interleukin-10 levels at baseline, week 4, 8, 12, 24 and 52 | baseline, 4, 8, 12, 24, and 52 weeks
  blood sample
interleukin-12P70 levels at baseline, week 4, 8, 12, 24 and 52 | baseline, 4, 8, 12, 24, and 52 weeks
  blood sample
interleukin-17 levels at baseline, week 4, 8, 12, 24 and 52 | baseline, 4, 8, 12, 24, and 52 weeks
  blood sample
Tumor necrosis factor -α levels at baseline, week 4, 8, 12, 24 and 52 | baseline, 4, 8, 12, 24, and 52 weeks
  blood sample
Interferon-γ levels at baseline, week 4, 8, 12, 24 and 52 | baseline, 4, 8, 12, 24, and 52 weeks
  blood sample
Interferon-α levels at baseline, week 4, 8, 12, 24 and 52 | baseline, 4, 8, 12, 24, and 52 weeks
  blood sample
interleukin-10 levels in tissue sample at baseline, week 12, 24 and 52 | baseline, 12, 24, and 52 weeks
  Intestinal mucosal tissue sample
interleukin-17 levels in tissue sample at baseline, week 12, 24 and 52 | baseline, 12, 24, and 52 weeks
  Intestinal mucosal tissue sample
Tumor necrosis factor -α levels in tissue sample at baseline, week 12, 24 and 52 | baseline, 12, 24, and 52 weeks
  Intestinal mucosal tissue sample
acetyl choline levels at baseline, week 12, 24 and 52 | baseline, 12, 24, and 52 weeks
  Intestinal mucosal tissue sample
Inflammatory Bowel Disease Questionnaire Score at baseline, week 12, 24 and 52 | baseline, 12, 24, and 52 weeks
  The range of Inflammatory Bowel Disease Questionnaire Score is 32-224, and higher scores mean worse outcome.
Gut metabolites profile at baseline, week 12, 24, and 52 | baseline, 12, 24, and 52 weeks
  fecal sample metabolites analysis
Gut microbiota profile at baseline, week 12, 24, and 52 | baseline, 12, 24, and 52 weeks
  fecal sample microbiota analysis
autonomic profile characteristics | baseline, 4, 8, 12, 24, and 36 weeks
  heart rate variability indicating sympathetic and parasympathetic activity
Hospital Anxiety and Depression scale score | baseline, 12, 24, and 52 weeks
  anxious depression. The range of Hospital Anxiety and Depression scale score is 0-21, and higher scores mean worse outcome.
Functional magnetic resonance imaging | baseline and 24 weeks
  blood oxygen level dependent，BOLD-fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Kaichun Wu, PhD, Study Chair — Air Force Military Medical University, China
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China